CLINICAL TRIAL: NCT06145958
Title: A Translational Study of Samples From the Radiotherapy and Androgen Deprivation In Combination After Local Surgery (RADICALS) Prostate Cancer Trial to Identify Those Most Likely to Benefit From Androgen Deprivation With Salvage Radiotherapy
Brief Title: Radiotherapy and Androgen Deprivation In Combination After Local Surgery (RADICALS) Translational Study
Acronym: RADICALS-TR
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 159874; 329626 (Other: IRAS)
Record Dates: First submitted 2023-11-13; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: biomarker
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The primary purpose of this study is to collect fixed tumour material in the previous RADICALS intervention trial. Cases are those receiving therapy vs controls receiving standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No androgen deprivation: Those patients not given androgen deprivation therapy
- Short course androgen deprivation: Those patients given 6 months of androgen deprivation therapy
  Interventions: Drug: Luteinising Hormone-Releasing Factor Analogue
- Long course androgen deprivation: Those patients given 24 months of androgen deprivation therapy
  Interventions: Drug: Luteinising Hormone-Releasing Factor Analogue

INTERVENTIONS:
Drug: Luteinising Hormone-Releasing Factor Analogue — Androgen Deprivation Therapy
  Groups: Long course androgen deprivation; Short course androgen deprivation

SUMMARY:
The goal of this translational study is to test the use of biomarkers in salvage treatment for prostate cancer after a previous operation to remove the prostate. The main question it aims to answer is:

• Can a biomarker identify a group of patients most likely to benefit from androgen deprivation therapy in conjunction with salvage radiotherapy No new participants will be involved, but tumour samples will be acquired, for patients that gave their permission in the completed RADICALS RT and HD studies.

DETAILED DESCRIPTION:
Early prostate cancer represents a wide spectrum of disease. Indolent disease is unlikely to ever become symptomatic and treatment is needlessly morbid and costly. Aggressive disease warrants intensification of therapy. Current clinical methods are poor at discriminating these outcomes.

The RADICALS trial was the largest trial conducted to date in men requiring further curative treatment after an operation. It already defined the role for radiotherapy after surgery (prostatectomy). The standard of care is now for blood test (PSA) monitoring after prostatectomy with radiotherapy offered when the PSA rises. The role and duration of hormone treatment (androgen deprivation), given in combination with radiotherapy, remains less clear. Currently if androgen deprivation is to be given, the RADICALS data support the use of a 24-month course, but this entails a considerable burden of side-effects for patients. Pathological and biological markers are needed to identify those most likely to benefit from androgen deprivation.

In RADICALS-TR, the investigators will conduct translational analyses on the biopsy and prostatectomy specimens from the RADICALS trial. The investigators aim to identify prognostic features and biomarkers predictive of benefit from androgen therapy. The investigators will prioritise the refinement and validation of clinical biomarkers already close to clinical utilisation. In this way it is hoped that findings can rapidly translate to stratified clinical trials and improved patient care.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

Diagnosis of nonmetastatic adenocarcinoma of the prostate Must have undergone radical prostatectomy Post-operative serum prostate-specific antigen (PSA) < 0.4 ng/mL No post-operative biochemical failure, defined as EITHER two consecutive rises in PSA and final PSA > 0.1 ng/mL OR three consecutive rises in PSA (for patients undergoing hormone therapy duration randomization)

Exclusion criteria:

Known distant metastases from prostate cancer PSA > 5 ng/mL at the time of hormone randomization (for patients undergoing hormone therapy duration randomization)

PATIENT CHARACTERISTICS:

* No other active malignancy likely to interfere with protocol treatment or follow-up.
* Consent has been given within the RADICALS (RT/HD) trial to translational research and follow up.

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

See Disease Characteristics Co-enrollment to other trials is permitted, providing this does not interfere with the outcome measures 5-α reductase inhibitors, soya, selenium, and vitamin E are acceptable non-trial therapies

Exclusion criteria:

Prior hormone therapy Bilateral orchidectomy Prior pelvic radiotherapy Neoadjuvant treatment Other concurrent therapies for prostate cancer (e.g., estrogens or cytotoxic chemotherapy) prior to disease progression

Ages: 18 Years to 99 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients were recruited to the RADICALS trial at one of two points:
  RT - after surgery for prostate cancer, possessing one or a number of higher risk features for subsequent relapse. These patients were randomised to either immediate radiotherapy or deferred until the point of biochemical relapse.
  HD - at the point of intiation of radiotherapy in the adjuvant or salvage setting. These patients were randomised to a number of different androgen deprivation durations (as detailed above in the cohort descriptions).
Sampling Method: Non-Probability Sample
Enrollment: 2585 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from Distant Metastases | Up to 12 years
  The absence of prostate cancer metastases

SECONDARY OUTCOMES:
Overall survival | Up to 12 years
  Freedom from death from any cause
Disease Specific Survival | Up to 12 years
  Freedom from prostate cancer specific death
Freedom from treatment failure | Up to 12 years
  Freedom from PSA progression whilst receiving androgen deprivation therapy
Clinical Progression Free survival | Up to 12 years
  Clinical progression of prostate cancer or initiation of non-protocol hormone therapy or death from prostate cancer.
Non protocol hormone therapy | Up to 12 years
  Initiation of hormone therapy other than that randomised.
Freedom from biochemical progression | Up to 12 years
  Where a biochemical progression event is defined as a PSA level of ≥0.4ng/ml following radiotherapy or a PSA level of > 2.0ng/ml regardless of prior radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Fittall, BMBCh PhD, Principal Investigator — UCL

IPD SHARING:
Plan to Share IPD: No
On request - clinical outcome data is available from the RADICALS trial team.